CLINICAL TRIAL: NCT02182271
Title: Safety, Tolerance, and Pharmacokinetics of Single Oral Doses of 5 mg, 20 mg, 60 mg, 150 mg, 300 mg, 600 mg, 1000 mg, and 1500 mg BI 201335 ZW (PEG 400/TRIS/Water Solution) in Healthy Male Subjects, in a Randomised Double Blind, Placebo Controlled Rising Dose Study, Followed With an Open-label Intra-subject Two-stage Crossover Pilot Bioavailability Comparison of 600 mg BI 201335 ZW in a PEG 400/TRIS/Water Solution Co-administered With Food
Brief Title: Single Rising Dose Study of BI 201335 ZW in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.1
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 201335 ZW - single rising dose (Experimental)
  Interventions: Drug: BI 201335 ZW - single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 201335 ZW - single rising dose
  Arms: BI 201335 ZW - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the current study is to investigate safety, tolerability, and pharmacokinetics of BI 201335 ZW following administration of single rising doses from 5 mg to 1500 mg. In addition Two stage intra-subject bioavailability comparison of 600 mg BI 201335 ZW as a liquid formulation given with and without food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria based upon a complete medical history, including the physical examination, vital signs ((blood pressure (BP), pulse rate (HR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and Age ≤55 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation
* Willingness to abstain from alcohol from screening period until conclusion visit

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders, including a clinical history of viral hepatitis, or serological evidence of active Hepatitis B or Hepatitis C infection
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range and of clinical relevance
* History of any familial bleeding disorder

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2004-10; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline, day 3 of each treatment period, within 8 days after last administration
Number of patients with clinically significant changes in vital signs | Baseline, day 1-3 of each treatment period, within 8 days after last administration
Number of patients with clinically significant changes in 12-lead ECG (electrocardiogram) | Baseline, day 1, 2 in treatment period, within 8 days after last administration
Number of patients with abnormal changes in laboratory parameters | Baseline, day 1-3 of each treatment period, within 8 days after last administration
Number of patients with adverse events | up to 13 days
Assessment of tolerability by investigator on a 4-point scale | on day 3 of each treatment period

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
tmax (time from dosing to maximum concentration) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
λz (terminal elimination rate constant in plasma) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
t1/2 (terminal half-life of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
MRTpo (Mean residence time of the analyte in the body after oral administration) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
CL/F (apparent clearance of the analyte in the plasma after oral administration) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 15, 24, 30, 36 and 48 hours post-dose